CLINICAL TRIAL: NCT04181983
Title: Personalized Exercise Programs for Older Adults - a Digital User-friendly Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Zinman College of Physical Education and Sports Sciences (Other)
Responsible Party: Principal Investigator, Jacobs Jeremy, Associate Professor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: JMJYN-HMO-CTIL
Record Dates: First submitted 2019-10-27; First posted 2019-12-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Healthy Older Adults; Exercise
Keywords: Home-based personalized exercise program; Smart phone application
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Personalized exercise program (Experimental): A home-based personalized exercise program using a smartphone app
  Interventions: Other: Personalized exercise program
- Active Control WHO guidelines (Active Comparator): A standard exercise program based upon WHO guidelines
  Interventions: Other: WHO exercise guidelines
- Control (No Intervention): No exercise program

INTERVENTIONS:
Other: Personalized exercise program — Home-based personalized exercise program using a smart phone app
  Arms: Personalized exercise program
Other: WHO exercise guidelines — Standard exercise counselling according to WHO guidelines
  Arms: Active Control WHO guidelines

SUMMARY:
Scientific Background:

Despite the known health benefits of exercising during old age, older people remain highly sedentary. Official exercise guidelines aimed specifically at older people focus primarily on aerobic activity, and tend to be over generalized.There is need for personalized exercise programs, which account for the increasing variability in measures of fitness and mobility with advancing age, and offer exercises aimed at improving balance, strength, flexibility and aerobic fitness, and which can be performed at home. Advancing smartphone technology provides tools which might help address this important area of public health.

Study Aims:

To develop a novel digital smartphone app, which enables assessment of fitness components, and provides personalized comprehensive exercise programs which update at regular intervals according to changes in fitness levels.

Methodology:

A prospective interventional randomized control study involving 360 people aged ≥65 living at home/ sheltered living. Stage 1 will include selecting exercise and fitness tests, developing a smartphone app for self-assessment of these tests, and designing exercise programs to meet specific capabilities. A pilot study (n=60) will validate results from the app compared to standard laboratory tests, before finalizing the study platform, and will create a platform for matching exercise programs to levels of fitness. At Stage 2 - the main study - participants (n=300) will be randomly assigned to the intervention group (personalized updating exercise program via the app), an active control group (receiving World Health Organization (WHO) exercise guidelines), or control group (no intervention). Using the app for assessment, all participants will be tested during stage 2 at T0 (baseline), T1 (6 week) T2 (12 weeks), and during Stage 3 follow-up at T3 (18 weeks) and T4 (24 weeks).

Novelty and Applicability:

This innovative technology will enable older people to test their fitness level, and receive a personalized exercise program based on their current ability and preferences, which changes over time according to their progress. The program will be presented as photos and short videos, available on their smartphones, or easily transferable to computer or television (TV) screens.

DETAILED DESCRIPTION:
1.1 Scientific Background

Although the health benefits of exercise among the elderly are accepted, there is a need for greater accuracy in assessment of a wide range of fitness and mobility parameters, in order to provide a comprehensive exercise program delivered in the home environment. Advances in smartphone technology may provide useful tools to help address this important area of public health.

1.2 Research Objectives

Aim: 1) To examine whether an individually prescribed personalized comprehensive physical activity program performed at home, based on individual motor and physical evaluation, performed by a standard smartphone at home, is more effective than accepted standardized recommendations from the World Health Organization for physical activity, among people aged 65 years and above. The prescribed program will include colorful, clear pictures and videos of various exercises, presented in a user-friendly manner on the user's smartphone, TV or computer screen.

Aim: 2) To enable the personalized exercise program to be updated (by the study exercise specialists), according to the changes in level of fitness, as measured by home testing using the smartphone.

Aim: 3) The ultimate goal of the program is to improve health of older people by increasing the level of physical activity in a safe, enjoyable and effective manner.

1.3 Research Design and Methods

We will employ an interventional, prospective randomized control study.

Ethical Approval: The study has been approved by the Hadassah Hospital Ethics Committee.

Participants:The study population will include a total of 360 community dwelling adults aged ≥65 years, without significant cognitive impairment, (60 adults in the Pilot Study, and a subsequent 300 adults in the Phase II main study).

Recruitment: Recruitment will be by flyers and lectures by the study PI's, at local elderly clubs, day centers, and independent living facilities (retirement homes).

Informed Consent: Informed consent will be attained following a detailed explanation given by the study physician experienced in geriatrics/exercise medicine (either the PI Prof Jacobs or Co Investigator-to be announced closer to the study initiation) concerning study details and any possible medical complications caused either directly (e.g. risk of falls and fractures, musculoskeletal pains, strained ligaments) or secondary to the exercise programs (e.g. cardiac arrhythmias or angina).

Study Procedure and design of research tools:

A. Phase I: Preliminary preparations and a pilot study:

1. Designing the tests.
2. Developing a dedicated digital app of the selected tests: 'Montfort Brain Monitor Ltd' will provide an app to enable measurement of the test battery using the mobile phone. Following testing using the smartphone at home, data will be remotely uploaded to the Montfort data bank for subsequent analysis.
3. Developing the Exercise Program: The photos and videos of the exercises will be presented in a user-friendly manner on the user's smartphone, TV or computer screen. Throughout the study period, participants will receive regular notifications via the smartphone, reminding them to exercise.
4. Pilot Study: Validation of the study instrument: Older adults (n=60), from the Netanya area (close to Wingate College) will be recruited for the pilot study. They will be tested using both the smartphone app as well as state of art laboratory tests, will be given an exercise program installed on their phone for performing at home, and will be tested again after 6 weeks of exercise.
5. Preparations for the main study: At this point, a study app will be finalized for running the smartphone app tests + running the matched exercise programs (provided individually by the research exercise specialists), and uploading data to the remote data bank for subsequent analysis.

B. Phase II: Main Study lasting 12 weeks:

Study participants (n=300) from day care centers, elderly clubs, retirement villages, etc., will be randomly assigned to 3 groups:

1. The experimental group: (n=100). Intervention-Personalized exercise program focusing upon Balance/Upper limb/shoulder flexibility and strength.
2. An active control group: (n=100). All participants in this group will receive exercise counseling and asked to exercise according to the official general guidelines published by the World Health Organization.
3. A control group: (n=100). Advised to continue their normal routine, and if interested, will be able use the smart app exercise program after the completion of the main study.

Participants from all groups will be tested individually by the tests app before (T0), after 6 weeks (T1), and after 3 months (T2).

C. Phase III: Follow-up:

The experimental group and the active control group will be re-assessed 6 weeks (T3) and 3 months (T4) following the termination of Phase II. The control group will get the treatment at that point, if they so desire.

Sample Size and Power Analysis: Statistical power was calculated using G * Power. Based on a 2-way ANOVA (3 groups X 5 tests) with repeated measures on the tests factor, 100 participants in each subgroup enable detecting group differences in statistical power of >99% for a moderate (Cohen's f = .25) and large (Cohen's f = .4) effect size. In addition, the statistical power for detecting differences between repeated measures, and in the interaction between groups in the repeated measures is higher than 99% in the moderate effect size as well as in the high effect size.

D. Additional Data Collection:

1. Sociodemographic data
2. Self-reported medical diagnosis and health related variables, Frailty Index
3. Level of physical activity
4. Mini-Cog test validated Hebrew version
5. Geriatric depression score (short 5 item validated Hebrew version )
6. Quality of life assessment ( Short Form-36, validated Hebrew version)

Study hypotheses

1. Participants in the experimental group (Personalized Balance/strength/flexibility exercise programs) will show greater improvement than participants with similar profiles in the active-control or control group.
2. Participants in the experimental group will adhere more to the exercise regime than participants in the active control group, thus will exhibit significantly more physical and motor improvements.
3. Both the experimental group and the active control group will gain more improvements in fitness than the non-active control.

Statistics: the selected digital tests for assessing the fitness components are to be determined in the first study phase. It is likely that a two-way Analysis of Variance (ANOVA, 3 groups X 5 measurements) with repeated measures on the measurements factor will be applied in most tests. Fisher Least Significant Difference will be used for post-hoc analyses. Significance level for all statistical tests will be set at alpha = .05.

1.4 Equipment and Films of exercises: The new exercises created for the current study will be photographed and/or filmed for video at the laboratory of education technology at the Wingate College.

Laboratory testing:

In order to establish the validity of the new dedicated mobile phone tests, participants of the pilot study will be tested on gold standard measurements at the biomechanical, physiological and motor control laboratories at the Wingate College. The laboratories are equipped with the following devices: Vicon Motion Capture Systems for 3D motion analysis (gait analysis and postural control), Biodex Medical Systems for isokinetic force measurements (strength of upper and lower extremities), motorized treadmill -Woodway, Germany (cardiovascular fitness - predicted VO2), and Balance Tutor (postural control, static and dynamic balance).

ELIGIBILITY:
Inclusion Criteria (all must be positive for inclusion)

* Living place: Home or Independent Living
* Fluent Hebrew speaker
* Ambulatory status: walks independently without help from another person
* Functional status: independent in dressing, toileting, grooming, washing, eating
* Smartphone user

Exclusion Criteria (any positive for exclusion)

* Cognitive decline <3/5 on Mini-Cog Score
* Hospitalization ( >24 hours) or Emergency Room referral in last 12 months due to unstable heart disease (congestive heart disease/rhythm disorder/ischemic heart disease/valvular heart disease) or neurological disease including balance or dizziness (cerebrovascular disease, vestibular disease, progressive neurological disease affecting gait or balance). (Information by self-report on direct questioning).
* High risk of falling (#): Any positive answer to one of the following questions: "Have you fallen over twice or more in the last year?", "Have you fallen and hurt yourself in the last year?", "Are you afraid that you might fall because of balance or walking problems?"
* Unwilling to provide consent.

(#) The identification of subjects at risk of falling will be based upon these three validated questions to identify and screen for increased risk of falling, used in community based exercise intervention and fall prevention studies:

1. Strategies to reduce injuries and develop confidence in elders (STRIDE): a cluster-randomized pragmatic trial of a multifactorial fall injury prevention strategy: design and methods. Bhasin S et al. Journal of Gerontology A Biological Science Medical Science,2018;73:1053-1061
2. Integration of balance and strength training into daily life activity to reduce rate of falls in older people (the Lifestyle integrated Functional Exercise (LiFE) study): randomized parallel study. Clemson L at al. British Medical Journal 2012;345:e547

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 239 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Balance | Changes in balance will be measured at the following points in time: Pilot study entry and 6 weeks later; Main study T0 (Baseline), T1 (6 weeks), T2 (12 weeks), T3 (18 weeks), T4 ( 24 weeks)
  1. Neutral stance eyes closed
  2. Right leg stance
  3. Left leg stance
  4. Tandem stance right
  5. Tandem stance left
  6. Tandem walk forward (10 steps)
  7. Tandem walk backward (10 steps)
  All the above will measure: range of acceleration in each direction (anterior-posterior, medio-lateral, superior-inferior) assessed in m/sec2
Balance | Changes in balance will be measured at the following points in time:Pilot study entry and 6 weeks later; Main study T0 (Baseline), T1 (6 weeks), T2 (12 weeks), T3 (18 weeks), T4 ( 24 weeks)
  Time-up-and-go:
  A composite measure of balance , which includes 1) the range of acceleration in each direction (anterior-posterior, medio-lateral, superior-inferior) assessed in m/sec2,2) the Number of steps taken (n), 3) Step length (cm).
Leg Strength | Changes in leg strength will be measured at the following points in time:Pilot study entry and 6 weeks later; Main study T0 (Baseline), T1 (6 weeks), T2 (12 weeks), T3 (18 weeks), T4 ( 24 weeks)
  Sit-to-stand
  A composite measure of leg strength based upon measurement of number of repetitions in 30 sec (n), and the acceleration range which will be measured in m/sec2
Upper extremities flexibility | Changes in upper extremities flexibility will be measured at the following points in time:Pilot study entry and 6 weeks later; Main study T0 (Baseline), T1 (6 weeks), T2 (12 weeks), T3 (18 weeks), T4 ( 24 weeks)
  1. Rotate torso to right
  2. Rotate torso to left
  3. Right arm flexion
  4. Right arm extension
  5. Right arm abduction
  6. Right arm to left shoulder at 90◦
  7. Right arm back folded
  8. Left arm flexion
  9. Left arm extension
  10. Left arm abduction
  11. Left arm to left shoulder at 90◦
  12. Left arm back folded
  The above tests are assessed by angle between arm and the horizon.
Upper extremities strength | Changes in upper extremities strength will be measured at the following points in time:Pilot study entry and 6 weeks later; Main study T0 (Baseline), T1 (6 weeks), T2 (12 weeks), T3 (18 weeks), T4 ( 24 weeks)
  1. Lifting right arm forward 20 times
  2. Lifting left arm forward 20 times
  3. Lifting right arm to the side 20 times
  4. Lifting left arm to the side 20 times
  For the above tests the range of acceleration will be assessed in m/sec2.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy M Jacobs, MBBS BSc, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah medical Organization, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Netz Y, Argov E, Yekutieli Z, Ayalon M, Tchelet K, Ben-Sira D, Amar Y, Jacobs JM. Personalized multicomponent exercise programs using smartphone technology among older people: protocol for a randomized controlled trial. BMC Geriatr. 2021 Oct 26;21(1):605. doi: 10.1186/s12877-021-02559-2. PMID 34702168